CLINICAL TRIAL: NCT00090259
Title: A Multi-center, Double-Blind, Randomized, Parallel Group Study to Evaluate the Effects of Two Different Doses of Losartan on Morbidity and Mortality in Patients With Symptomatic Heart Failure Intolerant of ACE Inhibitor Treatment
Brief Title: Study to Evaluate Potential Decrease in Hospitalization Events, Time Between Events, and Increasing Longevity in Patients With Symptomatic Heart Failure (0954-948)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-948; 2004_004
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Results first posted 2010-08-02 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Losartan 50 mg (Experimental): 50-mg losartan tablet administered daily with 1 tablet of 100-mg losartan placebo beginning Week 1 and continuing to end of study (up to 4 years)
  Interventions: Drug: Losartan 50 mg
- Losartan 150 mg (Experimental): Titrated losartan administration up to daily 150-mg losartan: Week 1, daily 50-mg losartan tablet coadministered with 100-mg losartan placebo; Week 2, daily 50-mg losartan placebo coadministered with 100-mg losartan; Week 3 to end of study (up to 4 years), daily 50-mg losartan tablet coadministered with 100-mg losartan
  Interventions: Drug: Losartan 150 mg

INTERVENTIONS:
Drug: Losartan 50 mg — 50-mg losartan oral tablet
  Other Names: Losartan potassium
  Arms: Losartan 50 mg
Drug: Losartan 150 mg — 100-mg losartan oral tablet + 50-mg losartan oral tablet
  Other Names: Losartan potassium
  Arms: Losartan 150 mg

SUMMARY:
This is a multicenter study to evaluate potential decrease in hospitalization events and time between events and increasing longevity in patients with symptomatic congestive heart failure and intolerant of first-line medication for heart failure. This study will evaluate if higher doses of the investigational drug given daily will be superior to the lower dose of the same investigational drug given daily.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure with known or recently diagnosed intolerance of treatment with first-line medication for heart failure
* May or may not be receiving an alternative and/or additional drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3834 (Actual)
Dates: Start 2001-12-19 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upshaw JN, Konstam MA, Klaveren Dv, Noubary F, Huggins GS, Kent DM. Multistate Model to Predict Heart Failure Hospitalizations and All-Cause Mortality in Outpatients With Heart Failure With Reduced Ejection Fraction: Model Derivation and External Validation. Circ Heart Fail. 2016 Aug;9(8):e003146. doi: 10.1161/CIRCHEARTFAILURE.116.003146. PMID 27514751
- [Derived] Rossignol P, Girerd N, Gregory D, Massaro J, Konstam MA, Zannad F. Increased visit-to-visit blood pressure variability is associated with worse cardiovascular outcomes in low ejection fraction heart failure patients: Insights from the HEAAL study. Int J Cardiol. 2015;187:183-9. doi: 10.1016/j.ijcard.2015.03.169. Epub 2015 Mar 17. PMID 25828348
- [Derived] Kiernan MS, Gregory D, Sarnak MJ, Rossignol P, Massaro J, Kociol R, Zannad F, Konstam MA. Early and late effects of high- versus low-dose angiotensin receptor blockade on renal function and outcomes in patients with chronic heart failure. JACC Heart Fail. 2015 Mar;3(3):214-23. doi: 10.1016/j.jchf.2014.11.004. PMID 25742759
- [Derived] Konstam MA, Neaton JD, Dickstein K, Drexler H, Komajda M, Martinez FA, Riegger GA, Malbecq W, Smith RD, Guptha S, Poole-Wilson PA; HEAAL Investigators. Effects of high-dose versus low-dose losartan on clinical outcomes in patients with heart failure (HEAAL study): a randomised, double-blind trial. Lancet. 2009 Nov 28;374(9704):1840-8. doi: 10.1016/S0140-6736(09)61913-9. Epub 2009 Nov 16. PMID 19922995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: Nov-2001. Last patient out: May-2009. 255 sites in 30 countries participated (Peru , Chile, Columbia, Mexico, Brazil, Belgium, Croatia, France, Germany, Greece, Holland, Italy, Norway, Poland, Russia, Slovenia, Spain, Turkey, UK, Egypt, Lebanon, Morocco, S. Africa, China, Hong Kong, Korea, Malaysia, Philippines, Singapore, Taiwan)
Pre-assignment Details: Patients who were on a Angiotensin II Antagonist (AIIA) had the option to begin losartan treatment with open-label losartan 12.5 mg for one week followed by losartan 25 mg for one week and were subsequently randomized to losartan 50 mg or losartan 150 mg.
Period: Overall Study
Arm/Group | Losartan 50 mg | Losartan 150 mg
Started | 1913 | 1921
Completed | 1851 (Completed follow-up: 963 on drug, 223 off drug, & 665 at death (death was considered an endpoint)) | 1873 (Completed follow-up: 1005 on drug, 233 off drug,& 635 at death (death was considered an endpoint))
Not Completed | 62 | 48
Not completed — Lost to Follow-up | 30 | 26
Not completed — Withdrawal by Subject | 21 | 15
Not completed — Investigator site closed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan 50 mg | Losartan 150 mg | Total
Number analyzed (Participants) | 1913 | 1921 | 3834
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [19 to 95] | 64.4 [18 to 98] | 64.2 [18 to 98]
Age, Customized [Number; unit: participants]
  < 65 years of Age | 889 | 879 | 1768
  >=65 years of Age | 1024 | 1042 | 2066
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 560 | 583 | 1143
  Male | 1353 | 1338 | 2691
Angiotensin II antagonists [Number; unit: Participants]
  No | 456 | 438 | 894
  Yes | 1457 | 1483 | 2940
New York Heart Association (NYHA) functional status [Number; unit: Participants] — NYHA Class Symptoms
  I No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  II Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    I No symptoms | 2 | 1 | 3
    II Mild symptoms | 1330 | 1327 | 2657
    III Marked limitation | 569 | 583 | 1152
    IV Severe limitations | 12 | 10 | 22
Region [Number; unit: participants]
  Asia and Pacific Region | 391 | 390 | 781
  East Europe | 212 | 207 | 419
  Middle East and Africa | 97 | 97 | 194
  Latin America | 309 | 315 | 624
  West Europe | 904 | 912 | 1816
β - Blocker therapy [Number; unit: Participants]
  No | 543 | 533 | 1076
  Yes | 1370 | 1388 | 2758

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced One Component of the Composite Clinical Endpoint of All Cause Death or Hospitalization for Heart Failure
Time Frame: Entire follow-up (median = 4.7 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | Losartan 50 mg | Losartan 150 mg
Number analyzed (Participants) | 1913 | 1921
Participants | 889 | 828
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 150 mg; Test type: Superiority or Other; p = 0.027, Regression, Cox; Model terms: treatment, region and β-blocker use at randomization; Hazard Ratio (HR) = 0.899, 95% CI 2-sided [0.818 to 0.988] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on Losartan 150 mg compared to Losartan 50 mg

2. Secondary Outcome: Number of Participants That Experienced One Components of the Composite Clinical Endpoint of All Cause Death or Cardiovascular Hospitalization
Description: Cardiovascular hospitalization is defined as any hospitalization that may be attributed to a cardiovascular cause, including heart failure.
Time Frame: Entire follow-up (median = 4.7 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | Losartan 50 mg | Losartan 150 mg
Number analyzed (Participants) | 1913 | 1921
Participants | 1085 | 1037
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 150 mg; Test type: Superiority or Other; p = 0.068, Regression, Cox; Model terms: treatment, region and β-blocker use at randomization; Hazard Ratio (HR) = 0.924, 95% CI 2-sided [0.848 to 1.006] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on Losartan 150 mg compared to Losartan 50 mg

3. Secondary Outcome: Number of Participants That Died (Any Cause)
Time Frame: Entire follow-up (median = 4.7 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | Losartan 50 mg | Losartan 150 mg
Number analyzed (Participants) | 1913 | 1921
Participants | 665 | 635
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 150 mg; Test type: Superiority or Other; p = 0.235, Regression, Cox; Model terms: treatment, region and β-blocker use at randomization; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.840 to 1.044] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on Losartan 150 mg compared to Losartan 50 mg

4. Secondary Outcome: Number of Participants That Were Hospitalized for Heart Failure
Time Frame: Entire follow-up (median = 4.7 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | Losartan 50 mg | Losartan 150 mg
Number analyzed (Participants) | 1913 | 1921
Participants | 503 | 450
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 150 mg; Test type: Superiority or Other; p = 0.025, Regression, Cox; Model terms: treatment, region and β-blocker use at randomization; Hazard Ratio (HR) = 0.865, 95% CI 2-sided [0.762 to 0.982] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on Losartan 150 mg compared to Losartan 50 mg

5. Secondary Outcome: Number of Participants That Experienced Cardiovascular Hospitalization
Time Frame: Entire follow-up (median = 4.7 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | Losartan 50 mg | Losartan 150 mg
Number analyzed (Participants) | 1913 | 1921
Participants | 826 | 762
Statistical Analysis 1: Comparison: Losartan 50 mg vs Losartan 150 mg; Test type: Superiority or Other; p = 0.023, Regression, Cox; Model terms: treatment, region and β-blocker use at randomization; Hazard Ratio (HR) = 0.892, 95% CI 2-sided [0.808 to 0.984] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on Losartan 150 mg compared to Losartan 50 mg

ADVERSE EVENTS:
Time Frame: All adverse experiences that occurred during or up to 14 days after permanent or temporary discontinuation of the study treatment were included in the safety analyses. Per guidelines, endpoints were not reported as serious adverse experiences.
Description: In all adverse experience tables, an individual is counted only once for each system organ class (SOC) (e.g. gastrointestinal disorders) where he/she reported one or more adverse experiences. The Medical Dictionary of Regulatory Activities (MedDRA) Version 12.0 was used in the generation of all tables used in this document.
Arm/Group | Losartan 50 mg | Losartan 150 mg
Serious Adverse Events (participants affected / at risk) | 691/1913 | 710/1921
Other Adverse Events (participants affected / at risk) | 1358/1913 | 1394/1921
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan 50 mg (N=1913) | Losartan 150 mg (N=1921)
Acquired haemophilia with anti FVIII, XI, or XIII (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 19 | 24
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 2
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 6
Atrial flutter (Cardiac disorders) | 0 | 3
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 8 | 5
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 3
Hydrocele (Congenital, familial and genetic disorders) | 2 | 2
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 2 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 2 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 3 | 1
Hyperthyroidism (Endocrine disorders) | 5 | 0
Hypothyroidism (Endocrine disorders) | 1 | 4
Cataract (Eye disorders) | 13 | 7
Diabetic retinopathy (Eye disorders) | 0 | 2
Eye haemorrhage (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 1 | 0
Parophthalmia (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 3 | 0
Retinopathy (Eye disorders) | 2 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7
Abdominal strangulated hernia (Gastrointestinal disorders) | 2 | 2
Acute abdomen (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Aphagia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 4 | 3
Dental caries (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Diverticulum (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 4 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 4
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 2
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 5 | 7
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 7 | 12
Gastritis erosive (Gastrointestinal disorders) | 3 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 13
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Giant cell epulis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 3 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Ileus paralytic (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 18 | 11
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 6 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 4
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 7 | 6
Pancreatitis acute (Gastrointestinal disorders) | 5 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 3 | 2
Periodontitis (Gastrointestinal disorders) | 0 | 1
Peritoneal effusion (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 3 | 3
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 6
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 | 13
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Blood creatinine increased (General disorders) | 2 | 5
Blood glucose abnormal (General disorders) | 1 | 0
Blood glucose increased (General disorders) | 0 | 3
Blood potassium decreased (General disorders) | 0 | 1
Blood potassium increased (General disorders) | 2 | 3
Blood pressure increased (General disorders) | 1 | 0
Blood sodium decreased (General disorders) | 1 | 0
Blood urea increased (General disorders) | 0 | 2
Blood urine present (General disorders) | 0 | 1
Cardioactive drug level above therapeutic (General disorders) | 1 | 0
Cardioactive drug level increased (General disorders) | 0 | 1
Coagulation time abnormal (General disorders) | 0 | 1
Coagulation time prolonged (General disorders) | 0 | 1
International normalised ratio increased (General disorders) | 2 | 2
Prothrombin time prolonged (General disorders) | 0 | 1
Red blood cell count decreased (General disorders) | 0 | 1
Urine cytology abnormal (General disorders) | 1 | 0
Weight decreased (General disorders) | 3 | 3
Weight increased (General disorders) | 0 | 1
White blood cell count increased (General disorders) | 0 | 1
Asthenia (General disorders) | 3 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 5 | 9
Chills (General disorders) | 1 | 0
Drug interaction (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 2
Generalised oedema (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 2
Hernia obstructive (General disorders) | 0 | 4
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 1 | 0
Implant site inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 9 | 1
Necrosis (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 11 | 10
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Perforated ulcer (General disorders) | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 3
Sudden death (General disorders) | 1 | 1
Ulcer haemorrhage (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 3 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 3
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 12 | 11
Cholecystitis acute (Hepatobiliary disorders) | 6 | 3
Cholelithiasis (Hepatobiliary disorders) | 11 | 15
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 2
Anaphylactic shock (Immune system disorders) | 2 | 1
Behcet's syndrome (Immune system disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 0 | 3
Abscess limb (Infections and infestations) | 0 | 2
Anal abscess (Infections and infestations) | 0 | 3
Appendicitis (Infections and infestations) | 5 | 4
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bone tuberculosis (Infections and infestations) | 1 | 0
Borrelia infection (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 18 | 12
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 4 | 3
Carbuncle (Infections and infestations) | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 11 | 9
Clostridial infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colon gangrene (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 4
Device related infection (Infections and infestations) | 2 | 2
Diabetic foot infection (Infections and infestations) | 1 | 3
Diarrhoea infectious (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 3 | 3
Empyema (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 8 | 5
Escherichia sepsis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 17 | 19
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Granuloma inguinale (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 1
Impetigo (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 0 | 2
Infected skin ulcer (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 4 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 5 | 8
Lung infection (Infections and infestations) | 3 | 8
Necrotising fasciitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 2
Otitis media chronic (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Penile abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 88 | 72
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 4 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 3 | 0
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 2 | 0
Pyoderma (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 10 | 12
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 18 | 20
Septic shock (Infections and infestations) | 7 | 9
Sinusitis (Infections and infestations) | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 2
Sweat gland infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Tuberculosis bladder (Infections and infestations) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Urinary tract infection (Infections and infestations) | 18 | 16
Urosepsis (Immune system disorders) | 3 | 6
Vaginal abscess (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 2 | 3
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 6
Wound infection bacterial (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 6
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 2
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 4
Cataract operation complication (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 2
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 2 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 11 | 12
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 6
Femur fracture (Injury, poisoning and procedural complications) | 6 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gas poisoning (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 4 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 4
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 2
Medical device complication (Injury, poisoning and procedural complications) | 1 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 3
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 15 | 16
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 3
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Postoperative renal failure (Injury, poisoning and procedural complications) | 2 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 5 | 1
Rib fracture (Injury, poisoning and procedural complications) | 8 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 16 | 15
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 6 | 2
Diabetic foot (Metabolism and nutrition disorders) | 6 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 4 | 4
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 8
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Lipomatosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Articular disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosis tendinous (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 21
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 3
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 16
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Superficial spreading melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Brain stem syndrome (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 3
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 4
Convulsion (Nervous system disorders) | 2 | 5
Dementia (Nervous system disorders) | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 7
Dizziness postural (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 2
Facial palsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypercapnic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 3
Parkinsonism (Nervous system disorders) | 0 | 1
Phantom pain (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 2
Radicular syndrome (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 3 | 0
Spinal cord herniation (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 12 | 5
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 2
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 2
Alcoholism (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 3 | 2
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 3
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 2
Personality disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Reactive psychosis (Psychiatric disorders) | 2 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 1 | 1
Azotaemia (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 5 | 3
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 5
Hydronephrosis (Renal and urinary disorders) | 1 | 3
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0
Nephritis allergic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 33 | 43
Renal failure acute (Renal and urinary disorders) | 21 | 21
Renal failure chronic (Renal and urinary disorders) | 7 | 6
Renal impairment (Renal and urinary disorders) | 4 | 9
Renal mass (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 6 | 7
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 11
Breast mass (Reproductive system and breast disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0
Hydrometra (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1
Perineal fistula (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 2 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Testicular haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine disorder (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 26 | 28
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Nodular vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Diabetic macroangiopathy (Vascular disorders) | 0 | 2
Extremity necrosis (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 6 | 4
Haemorrhage (Vascular disorders) | 0 | 2
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 4 | 4
Hypovolaemic shock (Vascular disorders) | 5 | 2
Intermittent claudication (Vascular disorders) | 1 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 3
Shock haemorrhagic (Vascular disorders) | 5 | 0
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2
Varicose ulceration (Vascular disorders) | 1 | 2
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan 50 mg (N=1913) | Losartan 150 mg (N=1921)
Anaemia (Blood and lymphatic system disorders) | 78 | 108
Angina pectoris (Cardiac disorders) | 100 | 100
Atrial fibrillation (Cardiac disorders) | 123 | 130
Cardiac failure (Cardiac disorders) | 231 | 200
Cardiac failure congestive (Cardiac disorders) | 106 | 92
Diarrhoea (Gastrointestinal disorders) | 136 | 159
Gastritis (Gastrointestinal disorders) | 98 | 82
Blood creatinine increased (General disorders) | 163 | 285
Blood glucose increased (General disorders) | 153 | 154
Blood potassium increased (General disorders) | 111 | 161
Blood urea increased (General disorders) | 159 | 222
Blood uric acid increased (General disorders) | 150 | 167
Chest pain (General disorders) | 119 | 109
Bronchitis (Infections and infestations) | 231 | 222
Influenza (Infections and infestations) | 111 | 116
Nasopharyngitis (Infections and infestations) | 170 | 195
Upper respiratory tract infection (Infections and infestations) | 90 | 107
Urinary tract infection (Infections and infestations) | 119 | 119
Diabetes mellitus (Metabolism and nutrition disorders) | 160 | 160
Back pain (Musculoskeletal and connective tissue disorders) | 135 | 121
Dizziness (Nervous system disorders) | 254 | 245
Headache (Nervous system disorders) | 116 | 100
Renal failure (Renal and urinary disorders) | 95 | 132
Cough (Respiratory, thoracic and mediastinal disorders) | 179 | 170
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 166 | 152
Hypertension (Vascular disorders) | 147 | 123
Hypotension (Vascular disorders) | 127 | 178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.